CLINICAL TRIAL: NCT01556659
Title: Left Ventricular Thrombus Formation After Acute Myocardial Infarction - a Randomized Multi-center Trial Comparing Two Different Anti-thrombotic Regimens
Brief Title: LV Thrombus After Acute AMI: A Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: VU University of Amsterdam (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jan Piek, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-004265-32
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Thrombosis Mural Following Myocardial Infarction
Keywords: Left ventricular thrombus; Acute myocardial infarction; Anticoagulation
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin K antagonist + (No Intervention): Treatment with carbasalaatcalcium 100 mg/day, P2Y12 inhibitors (clopidogrel 1x 75mg, ticagrelor 2x 90 mg or prasugrel 1x 10mg/day) and vitamin K antagonist (acenocoumarol)
- vitamin K antagonist - (Active Comparator): Treatment with carbasalaatcalcium 100 mg/day, P2Y12 inhibitors (clopidogrel 1x 75mg, ticagrelor 2x 90 mg or prasugrel 1x 10mg/day)
  Interventions: Drug: Absence of vitamin K antagonist

INTERVENTIONS:
Drug: Absence of vitamin K antagonist — Dual anti-platelet therapy
  Other Names: warfarin
  Arms: vitamin K antagonist -

SUMMARY:
Left Ventricular (LV) thrombus formation is witnessed in at least 10% of patients with ST segment elevation myocardial infarction (STEMI). It is a feared complication since it might increase the risk of thrombo-embolic events, including stroke. Guidelines recommend vitamin K antagonist treatment in these patients. However patients with STEMI nowadays undergo primary percutaneous coronary intervention (PCI) with coronary stent placement and consequently require dual anti-platelet therapy (ascal and P2Y12 inhibitors) to prevent stent thrombosis. Consequently, STEMI patients with LV thrombus are currently treated with triple antithrombotic therapy (aspirin, P2Y12 inhibitors, e.g. clopidogrel (75 mg/d) and vitamin K antagonist). Patients treated with triple antithrombotic therapy are subject to a strongly increased bleeding risk with a yearly incidence of 3.7% for dual anti-platelet therapy as compared to 12% for triple antithrombotic therapy. About 10% of these bleedings are cerebral. The mortality of such haemorrhagic strokes is 25%. A recent retrospective analysis did not show any beneficial effects of addition of vitamin K antagonist to dual anti-platelet therapy to prevent stroke. If vitamin K antagonist-therapy could be omitted, morbidity and mortality due to post-PCI bleedings will decrease. Therefore, a randomized trial is warranted to address this issue.

Design: A multicenter, prospective, randomized, two non-inferiority trial. The objective of the study is to determine in a randomized fashion the risks and benefits of the addition of vitamin K antagonists to dual anti-platelet therapy or dual anti-platelet therapy in patients with PCI-treated STEMI and LV thrombus formation on baseline echocardiography or baseline Magnetic Resonance Imaging (MRI).

DETAILED DESCRIPTION:
Design: A multicenter, prospective, randomized, non-inferiority trial with blinded evaluation of endpoints

Objective: The objective of this study is to determine in a randomized fashion the risks as well as the benefits of the addition of vitamin K antagonists to dual anti-platelet therapy in patients with PCI-treated STEMI and LV thrombus formation

Patients: Patients with acute myocardial infarction treated with primary PCI and LV thrombus on baseline echocardiography or baseline Magnetic Resonance Imaging. (MRI)

Methods: After written informed consent has been obtained, echocardiography and MRI are performed between 7-12 days after PCI. When LV thrombus is present on baseline MRI, patients are randomized to

1. Triple antithrombotic therapy (aspirin (100 mg/d), thienopyridine class antiplatelet agent,) and vitamin K antagonist (goal INR is 2.0 to 3.0))
2. Dual anti-platelet therapy (aspirin (100mg/d) and thienopyridine class antiplatelet agent, e.g. clopidogrel (75 mg/d).

Primary Endpoint: Primary outcome is defined as the proportions of patients with new cerebral micro-infarcts at 6 months relative to baseline measured by MRI.

Secondary Endpoints: The secondary endpoints as assessed at 6 and 12 months are:

* the composite of vascular death, recurrent myocardial infarction, stroke or systemic embolism
* presence of new cerebral mirco-bleeds
* the occurrence of major and minor bleeding
* neurological status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Left Ventricular thrombus on echocardiography or routine Magnetic Resonance Imaging
* Ongoing treatment with dual antiplatelet therapy according to ESC/ACC-AHA guidelines at the time of randomization.

Exclusion Criteria:

* Younger than 18
* Clinically or hemodynamically unstable
* Treatment with vitamin K antagonist prior to PCI or other expected indication for vitamin K antagonist treatment (e.g. atrium fibrillation) within the next 6 months
* Previous stroke or transient ischemic attack
* Scheduled for major surgery (including Coronary Artery Bypass Grafting) during the course of the study
* Active bleeding or high risk for bleeding contraindicating treatment with vitamin K antagonists
* Contra-indication for vitamin K antagonist treatment
* Chronic treatment with NSAIDs or COX-2 inhibitors for more than 4 days per week anticipated to continue during the study
* Congenital cardiac disease
* Presence of supraventricular or ventricular arrhythmias
* Expected candidate for ICD implantation with the next 6 months
* Severe renal impairment (estimated CrCl calculated by Cockcroft-Gault equation 5 30mL/min)
* Known or symptomatic brain disease (such as brain tumor)
* Women who are pregnant.
* Any contraindication for Contrast-Enhanced Magnetic Resonance Imaging (such as pacemaker, cerebrovascular clips, known contrast allergy, claustrophobia)
* Follow-up impossible (for example no fixed abode)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
The proportions of patients with new cerebral micro-infarcts at 6 months relative to baseline measured by MRI. | 6 months relative to baseline
  Primary outcome is defined as the proportions of patients with new cerebral micro-infarcts at 6 months relative to baseline measured by Magnetic Resonance Imaging.

SECONDARY OUTCOMES:
The presence of new cerebral micro-bleeds assessed by MRI | At 6 months and 12 months relative to baseline
Occurrence of major and minor bleeding | At 6 and 12 months relative to baseline
Neurological status | At 6 and 12 months relative to baseline
Quality of life using a validated checklist | At 6 and 12 months relative to baseline
Composite of vascular death, recurrent myocardial infarction, stroke or systemic embolism | At 6 and 12 months relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Piek, Prof, Principal Investigator — PI
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided